CLINICAL TRIAL: NCT06062407
Title: Screening Diagnosis of Fall Risk After Stroke and Initial Intervention: A Functional Near-infrared Spectroscopy (fNIRs) Study
Brief Title: Screening Diagnosis of Fall Risk After Stroke and Initial Intervention: A fNIRs Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dingqun Bai, Director, Department of rehabilitation medicine, Principal Investigator, Clinical Professor, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2023-810
Record Dates: First submitted 2023-09-06; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stroke subjects without fall risk: The patient was diagnosed with a stroke with a berg score of not less than 40.
- Stroke subjects with fall risk: The patient was diagnosed with a stroke with a berg score of less than 40.
- Healthy subjects: No history of stroke with normal lower limb motor function and balance

SUMMARY:
This is a functional near infrared spectroscopy (fNIRs) study designed to screen for risk of falls after diagnosis of stroke and initial intervention.

DETAILED DESCRIPTION:
This was an initial screening and preliminary intervention study. Each subject underwent two models of simultaneous fNIRs-EEG testing during the sit-to-stand process, the first without any intervention and the second based on biofeedback (EMG feedback) during the sit-to-stand process. Initial screening of fall risk in post-stroke patients was performed by comparing differences in brain activation and brain network connectivity between patients and healthy subjects. Preliminary validation the effectiveness of the EMG feedback-based sitting and standing training for post-stroke patients by comparing the differences of brain activation, brain network connectivity, and electromyographic changes during the sit-to-stand process in the two models.

ELIGIBILITY:
Inclusion Criteria:

Stroke patients 1. Diagnosis of stroke confirmed by neuroimaging (CT or MRI) evaluation 2. 18-85 years old 3. Able to complete the sit-to-stand transition 4. Able to follow instructions to complete the trial 5. Patients who signed an informed consent form.

Healthy Subjects: 1. No abnormalities on cranial fMRI examination 2. 18-85 years old 3. Able to complete the sit-to-stand transition 4. Able to follow instructions to complete the trial 5. not taking medications. 6. Subjects who signed an informed consent form

Exclusion Criteria:

Stroke patients: 1. Inability to tolerate the test due to organic diseases 2. Serious mental illness that prevents them from cooperating with or tolerating the trial 3. Pregnant or lactating women 4. Had metal implants, a history of other neurological disorders, acute cardiopulmonary dysfunction.

Healthy Subjects: 1. Inability to tolerate the test due to organic diseases 2. Serious mental illness that prevents them from cooperating with or tolerating the trial. 3. Pregnant or lactating women 4. Had metal implants, a history of other neurological disorders, acute cardiopulmonary dysfunction

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with stroke in the inpatient ward of the Department of Rehabilitation Medicine, The First Affiliated Hospital of Chongqing Medical University.
  Healthy subjects recruited through the Department of Rehabilitation Medicine, The First Affiliated Hospital of Chongqing Medical University.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Preliminary screening of brain function biomarkers for fall risk in post-stroke patients | 1 day
  Comparison of differences in brain activation [HbO2 (mmol/L*mm)] between post-stroke patients with fall risk and healthy subjects
The brain functional effectiveness of the EMG feedback-based standing training | 1 day
  Comparison of the differences in brain activation [HbO2 (mmol/L*mm）] during the sit-to-stand process in the two models.
The neuromuscular activity of the EMG feedback-based standing training | 1 day
  Comparison of the differences in electromyographic changes [EMG (uv)] during the sit-to-stand process in the two models.

CONTACTS AND LOCATIONS:
Overall Officials: Dingqun Bai, Study Chair — The Department of Endocrinology, The First Affiliated Hospital of Chongqing Medical University
Locations (1):
- Department of Rehabilitation Medicine, the First Affiliated Hospital of Chongqing Medical University, Chongqing, China

REFERENCES:
- [Derived] Yang Z, Ye L, Yang L, Lu Q, Yu A, Bai D. Early screening of post-stroke fall risk: A simultaneous multimodal fNIRs-EMG study. CNS Neurosci Ther. 2024 Sep;30(9):e70041. doi: 10.1111/cns.70041. PMID 39315509